CLINICAL TRIAL: NCT06994221
Title: Assessment of Myocardial Fibrosis by 18F-FAPI/PET-CT in Patients With Myocardial Infarction-associated Ventricular Aneurysm
Brief Title: Fibrosis Assessment in Myocardial Infarction-associated Ventricular Aneurysm
Status: Recruiting | Type: Observational
Sponsor: RenJi Hospital (Other)
Responsible Party: Principal Investigator, Zhiguo Zou, Doctor, RenJi Hospital
Other Study IDs: EARLY-MYO FAPI-PET/CT
Record Dates: First submitted 2025-05-20; First posted 2025-05-29 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Acute Myocardial Infarction; Ventricular Aneurysm Following Acute Myocardial Infarction; Myocardial Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Acute myocardial infarction-associated ventricular aneurysm: Participants in this group are patients diagnosed with a ventricular aneurysm secondary to acute myocardial infarction (AMI). Diagnosis of AMI is based on clinical presentation, elevated cardiac biomarkers, ECG changes, and coronary angiogram. Ventricular aneurysm is mainly diagnosed by imaging modalities such as echocardiography and cardiovascular magnetic resonance (CMR).
  Interventions: Diagnostic Test: 18F FAPI-42 PET/CT scan
- Acute myocardial infarction without evidence of ventricular aneurysm: Participants in this group are patients diagnosed with AMI only. Diagnosis of AMI is based on clinical presentation, elevated cardiac biomarkers, ECG changes, and coronary angiogram. Echocardiography or CMR does not identify a ventricular aneurysm.
  Interventions: Diagnostic Test: 18F FAPI-42 PET/CT scan

INTERVENTIONS:
Diagnostic Test: 18F FAPI-42 PET/CT scan — During the hospital stay, participants will receive an 18F FAPI-42 PET/CT scan. 18F FAPI-42 is a new fibroblast activation protein (FAP)-specific tracer used for fibrosis imaging. PET/CT will be performed using the ultra-high-resolution digital PET/CT uEXPLORER (United Imaging, Shanghai, China)

SUMMARY:
The study will use 18F-FAPI PET/CT to study myocardial fibrosis in patients diagnosed with myocardial infarction-associated ventricular aneurysm (MI-VA). Participants will receive the PET/CT scan during hospital stay, as well as serial echocardiography and telephonic follow-ups. Analysed will focus on the characterization of myocardial fibrosis and its correlations with the clinical prognosis in the patients.

DETAILED DESCRIPTION:
The aim of this study is to investigate the temporal and spatial distribution of myocardial fibrosis in patients diagnosed with myocardial infarction-associated ventricular aneurysm using the novel fibroblast activation imaging tracer 18F FAPI-42 with PET/CT. This imaging modality allows for non-invasive visualization of activated fibroblasts, which are a key component of myocardial fibrotic remodeling after infarction.

The study is expected to enroll patients diagnosed with ventricular aneurysm secondary to acute myocardial infarction (AMI), who are hospitalized at Renji Hospital, Shanghai Jiao Tong University School of Medicine. The investigators expect to enroll 20 patients diagnosed with MI-VA and 10 AMI patients without evidence of ventricular aneurysm. With written informed consent, the investigators will review past medical records and document the medical history for each participant. During the hospital stay, participants will receive an 18F FAPI-42 PET/CT scan. FAPI uptake in the ventricular aneurysm and remote myocardium will be calculated as maximum standardized uptake value (SUVmax) and mean standardized uptake value (SUVmean). Correlation between SUVmax/SUVmean and critical markers of the disease progression, such as B-type natriuretic peptide (BNP) and cardiac troponin I (cTnI), will be analysed by Pearson or Spearman correlation coefficients. All participants will be followed for 1 year after enrolment, and serial echocardiography and telephonic follow-up will be performed. Major adverse cardiovascular events (MACE) will be recorded throughout the follow-up to reveal any predictive values of 18F-FAPI PET/C-assessed fibrosis for the patients with MI-VA.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-75 years old
* Diagnosed with STEMI or NSTEMI (ACC/AHA guidelines)
* Half male and half female
* Undergo CAG and PCI treatment;
* Receive either echocardiography or CMR to identify a ventricular aneurysm;
* Written informed consent

Exclusion Criteria:

* Patients under the age of 18 years old;
* Patients who are pregnant/breastfeeding;
* Patients who has a previous history of allergy to radio tracers.

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Enrolled patients are expected to be diagnosed with ventricular aneurysm secondary to acute myocardial infarction (AMI), and are hospitalized at Renji Hospital, Shanghai Jiao Tong University School of Medicine. The investigators expect to enroll 20 patients diagnosed with MI-VA and 10 AMI patients without evidence of ventricular aneurysm.
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
FAPI uptake (SUV max) | Day 1 after the PET/CT scan.
  FAPI uptake is assessed by drawing regions of interest (ROI), and determined as the maximal standard uptake value (SUVmax).
FAPI uptake (SUV mean) | Day 1 after the PET/CT scan.
  FAPI uptake is assessed by drawing regions of interest (ROI), and determined as the mean standard uptake value (SUVmean).

SECONDARY OUTCOMES:
Cardiac function assessed by echocardiography | Day 1 after the PET/CT scan, and at 1-month, 6-month and 1-year follow-ups
  Cadiac function is evaluated as left ventricular ejection fraction (LVEF, %) by echocardiography
The event rate of heart failure | From date of enrollment until the date of follow-ups at 1 month, 6 month and 1 year post discharge.
  The proportion (%) of participants who experience symptomatic heart failure. Heart failure is diagnosed based on symptoms such as shortness of breath and excess fluid, in the presence of a reduced LVEF (<60%) as assessed by echocardiography.

CONTACTS AND LOCATIONS:
Locations (1):
- Renji Hospital, Shanghai, China